CLINICAL TRIAL: NCT04377698
Title: 'A Comparison of Platelet Rich Fibrin & Mineralised Freezed Dried Bone Allograft to Radiographically Evaluate Healing Post Endodontic Surgery'- an In-vivo Study
Brief Title: PRF and Bone Graft in Endodontic Surgeries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Saraswati Dental College (Other)
Responsible Party: Principal Investigator, Madhur Garg, Principal Investigator, Saraswati Dental College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SDC/IRDC/2017/MDS-P/05
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Periapical; Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Platelet Rich Fibrin group(PRF) (Active Comparator): Following apicoectomy PRF gel was prepared and placed in the osseous defect followed by placement of PRF membrane
  Interventions: Biological: Platelet Rich Fibrin
- Freezed Dried Bone Allograft group(FDBA) (Active Comparator): Following apicoectomy FDBA graft were prepared and placed in the osseous defect followed by placement of PRF membrane
  Interventions: Biological: FDBA

INTERVENTIONS:
Biological: Platelet Rich Fibrin — regeneration, restoration or reconstitution of the lost periapical tissues of the tooth by using regenerative therapies that utilize growth factors and barrier membranes.
  Arms: Platelet Rich Fibrin group(PRF)
Biological: FDBA — regeneration, restoration or reconstitution of the lost periapical tissues of the tooth by using regenerative therapies that utilize growth factors and barrier membranes.
  Arms: Freezed Dried Bone Allograft group(FDBA)

SUMMARY:
AIM: The aim of this study was to compare and evaluate the radiographic healing in patients undergoing apical surgery, using Freeze dried mineralized bone allograft and Platelet-rich Fibrin. OBJECTIVES: To evaluate radiographic healing after periapical surgery using Freeze dried mineralized bone allograft. To evaluate radiographic healing after periapical surgery using Platelet rich Fibrin. To compare the radiographic healing after periapical surgery using Freeze dried mineralized bone allograft and Platelet rich Fibrin. Method: Patients were selected(according to the inclusion criteria) and randomly allocated to PRF and Bone Graft groups.Following apicoectomy PRF gel and FDBA graft were prepared and placed in the osseous defect followed by placement of PRF membrane for graft stabilization and flap closure. Radiographic follow up was done at 1st, 3rd, 6th and 12th months for evaluation of healing using Molven Criteria.

DETAILED DESCRIPTION:
The present study will be carried out to compare the post surgical healing of Platelet Rich Fibrin (PRF) & Mineralised freeze-dried bone allograft (FDBA) in the Department of Conservative Dentistry & Endodontics at Saraswati Dental College, Lucknow. The study will be commenced only after due permission and clearance from the Institutional Review Board and Ethical Committee.

Cases will be selected according to the inclusion criteria after obtaining informed consent from the parents. Patients will be diagnosed based on clinical signs & symptoms, intraoral & radiographic findings. A routine medical history followed by blood investigations will be part of the surgical protocol.

After meeting the above criteria the patients will be randomly assigned to either PRF group (Group-A) or Mineralised FDBA group (Group-B) After successful administration of Local Anaesthesia the surgical procedure will be carried out that will include reflection of a full thickness mucoperiosteal flap by sulcular incision and two relieving vertical incisions. Debridement of tissues at the defect site will be done followed by irrigation with sterile saline solution.

In Group-A patients :- 10ml of venous blood will be drawn from the patients by using a 18 gauge needle after selecting a suitable site for venipuncture. Blood will be collected in tubes without anticoagulant and immediately centrifuged at 3,000 rpm for 10min which will result in a fibrin clot containing the platelets located in the middle of the tube, between a layer of red blood cells at the bottom and acellular plasma at the top. This clot will be removed from the tube and the attached red blood cells will be scraped off and discarded.

PRF will be placed into the defect site and wound closure will be performed using appropriate sutures.

In Group-B patients :- Graft material i.e., Mineralised freeze-dried bone allograft (obtained from Tissue Bank, Tata Memorial Hospital) will be mixed with sterile saline solution, followed by careful placement into the defect site.

The flap will be then re-placed to its original position and sutured with appropriate sutures to ensure complete soft tissue coverage of the graft site.

Sutures will be removed after 7 days post-operatively. The cases will be followed up with clinical and radiographic examination and will be recalled at intervals of 3,6, and 9 months to assess the periapical area.

*Any changes in the plan of study will be made as in when necessary following which suitable statistical analysis will be used to analyse the result.

ELIGIBILITY:
Inclusion Criteria:

* Adult teeth with failed conventional endodontic therapy and a need for periapical root end surgery.
* Teeth with bony defect confined to periapical area.
* Adult individuals presenting a tooth with persisting periapical radiolucency.
* Adult individuals presenting a tooth with persistent fistula.
* Adult individuals presenting a tooth with persisting symptoms after orthograde re-treatment.

Exclusion Criteria:

• Patients with severe systemic disorder (i.e. uncontrolled diabetes, immunologic diseases, malignancy), thrombocytopenia or insufficient compliance.

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Change in radiographic healing of periapical tissue after Apicoectomy | Change from Baseline radiographic score at 1 month
  Two endodontists extraneous to the present study evaluated the radiographs post intervention and scored the healing according to Molven's scoring criteria for radiographic healing where 0 is representative of unsatisfactory healing and 3- complete healing
Change in radiographic healing of periapical tissue after Apicoectomy | Change from Baseline radiographic score at 3 months
  Two endodontists extraneous to the present study evaluated the radiographs post intervention and scored the healing according to Molven's scoring criteria for radiographic healing where 0 is representative of unsatisfactory healing and 3- complete healing
Change in radiographic healing of periapical tissue after Apicoectomy | Change from Baseline radiographic score at 6 months
  Two endodontists extraneous to the present study evaluated the radiographs post intervention and scored the healing according to Molven's scoring criteria for radiographic healing where 0 is representative of unsatisfactory healing and 3- complete healing
Change in radiographic healing of periapical tissue after Apicoectomy | Change from Baseline radiographic score at 12 months
  Two endodontists extraneous to the present study evaluated the radiographs post intervention and scored the healing according to Molven's scoring criteria for radiographic healing where 0 is representative of unsatisfactory healing and 3- complete healing

CONTACTS AND LOCATIONS:
Overall Officials: Madhur Garg, Principal Investigator — Saraswati Dental College
Locations (1):
- Madhur Garg, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No